CLINICAL TRIAL: NCT03011957
Title: Biomarkers for Muscle Function and Aging in Chronic HIV Infection
Acronym: MATCH
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Brigham and Women's Hospital (Other)
Responsible Party: Principal Investigator, Monty Montano, Director, Muscle and Aging Interventions, Brigham and Women's Hospital
Other Study IDs: 2014P002489
Record Dates: First submitted 2016-12-12; First posted 2017-01-06 (Estimated); Last update posted 2018-01-18 (Actual); Status verified 2018-01

CONDITIONS: HIV

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, muscle biopsy
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: HIV positive viral load < 200 copies/ml 50-65 years old CD4 > 350 cells/ml Male or Female
- Group 2: HIV negative 50-65 years old CD4 > 350 cells/ml Male or Female

SUMMARY:
MATCH is an observation study of HIV-infected adults on effective antiretroviral therapy (ART) and demographically matched uninfected adults to evaluate muscle and aging.

DETAILED DESCRIPTION:
MATCH is a non-randomized observational longitudinal study. We will recruit HIV infected adults (50 to 65 years old) and demographically matched uninfected control subjects to be followed for 4 years over the course of a 5 year study. The targeted age range of 50-65 is chosen to evaluate aging HIV infected individuals at risk for early frailty in the United States. All subjects will undergo blood draws and physical function assessment, and a subset will undergo a CT scan of muscle and will have a muscle biopsy taken.

A substudy will be performed on a subgroup of HIV-infected and HIV-uninfected men from the main cohort to measure daily physical activity by using an activity tracker.

ELIGIBILITY:
Inclusion Criteria:

Group 1: HIV positive subjects

* HIV positive
* English speaking
* 50-65 years old
* On Antiretroviral therapy and an HIV viral load below 200 copies/ml
* CD4 equal to or greater than 350 cells/mm3
* Postmenopausal (women)
* Lower extremity mobility sufficient to participate in functional assessment.

Group 2: HIV negative subjects Inclusion Criteria for Group 2 subjects

* English speaking
* 50-65 years old
* Negative for HIV (based on an HIV antibody test at Study Visit 1)
* Matched to Group 1 for sex (50% W, 50% M) and age (50 - 65yo)
* Postmenopausal (women)
* Lower extremity mobility sufficient to participate in functional assessment.

Exclusion Criteria:

Exclusion Criteria for Group 1 Subjects

* Acute or serious illness within 60 days prior to entry
* Use of pharmacologic doses of corticosteroids in the past 6 months.
* Use of anabolic therapy in the past 6 months.
* Lower extremity mobility insufficient to participate in functional assessment.
* Current use (last 30 days) of anticoagulants or known bleeding disorder.

Exclusion Criteria for Group 2 subjects

* Acute or serious illness within 60 days prior to entry
* Use of pharmacologic doses of corticosteroids in the past 6 months
* Use of anabolic therapy in the past 6 months
* Lower extremity mobility insufficient to participate in functional assessment
* Current use (last 30 days) of anticoagulants or known bleeding disorder.

Ages: 50 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Group 1: 66 HIV+ (both men and women), 50 through 65 years of age, on effective antiretroviral therapy (ART).
  Group 2: 94 HIV- (both men and women), 50 through 65 years of age.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2015-02; Primary Completion 2019-02 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
Inflammation at baseline and 3 years | 3 years
  Inflammation at baseline and yearly for 3 years will be assessed by measuring circulating levels of inflammatory cytokines (e.g., CRP, IL6) and soluble monocyte/macrophage biomarkers (e.g., sCD14, sC163). These multiple measurements will be aggregated to arrive at one composite inflammatory score. Outcome will be assessed in association with HIV status and physical function.

CONTACTS AND LOCATIONS:
Overall Officials: Monty A Montano, PhD, Principal Investigator — Brigham and Womens Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Only aggregate data will be made available through publication

REFERENCES:
- [Result] Tran T, Guardigni V, Pencina KM, Amato AA, Floyd M, Brawley B, Mozeleski B, McKinnon J, Woodbury E, Heckel E, Li Z, Storer T, Sax PE, Montano M. Atypical Skeletal Muscle Profiles in Human Immunodeficiency Virus-Infected Asymptomatic Middle-Aged Adults. Clin Infect Dis. 2018 Jun 1;66(12):1918-1927. doi: 10.1093/cid/cix1121. PMID 29293942